CLINICAL TRIAL: NCT06085573
Title: Precedex Intravenous Solution Special Investigation (Sedation of Non-intubated Pediatric Patients for Non-invasive Procedures and Tests)
Brief Title: A Study to Learn About the Study Medicine - Precedex in Children From Japan.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C0801044; NCT06085573 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sedation
Keywords: Precedex;; Dexmedetomidine Hydrochloride;; Sedation;; non-intubated;; pediatric;; non-invasive procedures and tests
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Dexmedetomidine Hydrochloride: Pediatric patients (1 month to < 18 years old) administered Precedex (Dexmedetomidine Hydrochloride) for "sedation of non-intubated pediatric patients for non-invasive procedures and tests"
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — <Sedation of non-invasive procedures and tests without intubation in pediatrics> For children aged 2 years or older, the usual dosage of dexmedetomidine is 12 μg/kg/hr given as a continuous intravenous infusion over 10 minutes (initial loading dose) followed by a maintenance dose of 1.5 μg/kg/hr (maintenance dose).
  For children aged 1 month to < 2 years old, the usual dosage of dexmedetomidine is 9 μg/kg/hr given as a continuous intravenous infusion over 10 minutes (initial loading dose) followed by a maintenance dose of 1.5 μg/kg/hr (maintenance dose).
  The infusion rate should be reduced according to patient's condition.
  Other Names: Precedex

SUMMARY:
The purpose of this study is to look at the safety of Precedex when it was used to calm children at procedures or tests under actual medical practice in Japan.

This study is seeking for children who are 1 month to less than 18 years old.

The patients are planned to be looked over:

* From the time of patient check before receiving Precedex
* To 1 hour after the completion or stop of using Precedex.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (1 month to < 18 years old) administered Precedex for "sedation of non-intubated pediatric patients for non-invasive procedures and tests"

Exclusion Criteria:

* No exclusion criteria is set out in this study.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients (1 month to < 18 years old) administered Precedex for "sedation of non-intubated pediatric patients for non-invasive procedures and tests"
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse drug reactions (ADRs) | From the time of patient assessment before the start of administration of Precedex to 1 hour after the completion or discontinuation of administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Toykyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0801044